CLINICAL TRIAL: NCT03263949
Title: Predicting Ventricular Tachyarrhythmias Following Acute ST Elevation Myocardial Infarction
Acronym: PREDICT-VT
Status: Completed | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Igor Mrdovic, Professor, Clinical Centre of Serbia
Other Study IDs: 1533/17
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Risk Stratification
Keywords: risk prediction; ventricular arrhythmia; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic — For the analysis of myocardial function, conventional 2D echocardiography and tissue doppler will be used. For the evaluation of myocardial mechanics, 2D speckle tracking, strain, strain rate and mechanical dispersion will be obtained.

SUMMARY:
Predict-VT is an investigator-initiated, prospective, observational clinical trial. Four hundred patients with ST elevation acute myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI) will be included. The primary end point is a composite of ventricular tachyarrhythmia (VTA) and sudden cardiac death (SCD). VTAs will be recorded using continuous electrocardiographic (ECG) monitoring in the coronary unit for the first 72 hours, standard ECG and ECG holter monitoring. For the analysis of myocardial function, conventional 2D echocardiography and tissue doppler will be used. For the evaluation of myocardial mechanics, 2D speckle tracking, strain, strain rate and mechanical dispersion will be obtained. Important clinical, laboratory and angiographic variables will also be examined. Patients will be followed-up at 40 days and 1 year. The optimal VTA prediction model will be constructed using logistic regression and bootstrap models. Patients who experience primary end point should undergo secondary SCD prevention using implantable cardioverter defibrillator (ICD). Patients with left ventricular ejection fraction (LVEF) < 35%, 40 days post acute myocardial infarction (AMI), will be candidates for primary SCD prevention.

DETAILED DESCRIPTION:
Study design Predict-VT is an investigator-initiated, prospective, open-label, single-center clinical trial. The research protocol has been approved by the Ethics Committee of the Clinical Center of Serbia. All participants will have to provide their informed consent in writing. The trial design will ensure that all participants abide by good clinical practice and the ethical principles of the Declaration of Helsinki II.

Study population The study will include at least 400 patients with acute myocardial infarction with ST elevation (STEMI) who are elgible for treatment with primary percutaneous coronary intervention (PPCI) within 12 hours from the onset of symptoms. Enrollment started on January 2017 . Recruitment will continue until 400 patients have been randomized. The end of the recruitment period is planned for January 2021. The trial will continue until all available survivors have been followed for at least 1 year.

Objectives, end points and definitions The primary objective of PREDICT-VT trial is to test the hypothesis that the occurrence of ventricular tachyarrhythmias (VTA) and sudden cardiac death (SCD) is predictable with acceptable accuracy among STEMI patients undergoing PPCI. Therefore, the PREDICT-VT specified primary end point is the analysis of independent predictors of VTA and SCD in a period of 3-40 days following STEMI. The second objective of the study is the stratification of risk for VTA by constructing optimal predictive models and defining the classes of risk. The third objective of the study is a validation of the model using an independent sample of patients. The study's subanalyses will include: a. Analysis of the significance of non-sustained VTA lasting <30 seconds for the prognosis of patients with STEMI, b. Importance of frequent ventricular premature beats and/or emerging atrial fibrillation for the prognosis of patients and the emergence of SCD, c. Definition of risk factors for the occurrence of VTA in the subgroup of patients with preserved left ventricular ejection fraction (LVEF), considering that more than half of the SCD victims have preserved LVEF.

Noninvasive and invasive assessment A 24-hour ECG Holter monitoring will be performed in the period of 5 ± 2 days after STEMI.

Echocardiographic examination on Vivid E9 (General Electric) echocardiographic device will be performed 5 ± 2 days after STEMI and repeated after 50 ± 10 days. Standard echocardiographic methods of M-mode, 2D, color, pulse, continuous doppler, tissue doppler and 2D speckle tracking will be used. The analysis will include the parameters of systolic and diastolic functions and myocardial mechanics in accordance with the latest recommendations of the European / American Echocardiographic Association.

The following angiographic variables will be analyzed: significant coronary artery stenosis -localization and number, number of diseased coronary vessels, length of stenosis, type of stenosis, coronary flow before and after the intervention, type and number of implanted stents.

Patients will be followed-up after discharge from hospital for the occurrence of specified end points at 40 days and 1 year after enrollment by scheduled telephone interviews and outpatient visits. An independent Clinical Event Committee, composed of 3 cardiologists will review and adjudicate the occurrence of each suspected clinical end point.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* willing consent in writing
* undergoing primary PCI for STEMI

Exclusion Criteria:

* cardiogenic shock at admission,
* noncardiac conditions that could interfere with compliance with the protocol,
* coexisting conditions associated with a limited life expectancy in the follow-up period.
* Prior documented arrhythmias like atrial fibrillation or ventricular tachyarrhythmias,
* Permanent pacemaker implanted,
* Previous haemodynamically significant valvular abnormalities,
* Chest wall deformities disabling adequate echocardiographic examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 600 patients with acute myocardial infarction (AMI) with ST elevation (STEMI) who are eligible for treatment with primary percutaneous coronary intervention (PPCI) within 12 hours from the onset of symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Composite of ventricular tachyarrhythmias and sudden cardiac death | 3-40 days after STEMI
  Analysis of independent predictors of ventricular tachyarrhythmias and sudden cardiac death in a period of 3-40 days following STEMI. Predictors will be identified from clinical, laboratory, echocardiographic, angiographic and procedural variables collected in the study database, using statistical methods of univariable logistic regression and Cox proportional hazard model. Statistical methods of multivariable logistic regression, bootstrapping and receiver operating characteristic curve analysis will be used for the identification of independent predictors of outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Mrdovic, Principal Investigator — Clinical Centre of Serbia
Locations (1):
- Clinical Centre of Serbia, Emergency Hospital, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No